CLINICAL TRIAL: NCT00967122
Title: The Effect of Lap Band Adjustment on Satiety Peptides
Brief Title: Band Holiday Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Principal Investigator, Heekoung A Youn, Research coordinator, NYU Langone Health
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NYUSWLP-BH
Record Dates: First submitted 2009-08-25; First posted 2009-08-27 (Estimated); Last update posted 2012-09-27 (Estimated); Status verified 2012-09

CONDITIONS: Famine
Keywords: adjustment, hunger; Hunger/satiety changes before and after gastric band adjustment
MeSH Terms: interventions — Specimen Handling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- No Arm (No Intervention)
  Interventions: Procedure: Band adjustment and specimen collection

INTERVENTIONS:
Procedure: Band adjustment and specimen collection — Clinical evaluation and sample collection before and after band adjustment

SUMMARY:
AIMS: Our aims are to measure BMI and plasma concentrations of representative hormones before and after a band holiday, in addition to surveying hunger/satiety and behavior changes.

DETAILED DESCRIPTION:
AIMS: Our aims are to measure BMI and plasma concentrations of representative hormones before and after a band holiday, in addition to surveying hunger/satiety and behavior changes.

Materials and Methods:

Adults ≥ 18 years of age who previously underwent LAGB at New York University Medical Center and have lost sufficient excess body weight and agree to have their band temporarily loosened for a 2 week period will be invited by the health care provider to participate. Patients of both genders and all races are eligible for participation. Patients will need to consent to complete a questionnaire and to have blood drawn when the band is loosened and refilled. Patients will only be excluded if they are not willing to have their band loosened or if they will not present for follow-up.

Sample size:

For this pilot program we plan to enroll 15 patients. Since patients will serve as their own controls before and after meals as well as before and after band adjustments, we anticipate adequate power to assess for significant variations.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years of age
* who previously underwent LAGB at New York University Medical Center and have lost sufficient excess body weight and
* agree to have their band temporarily loosened for a 2 week period will be invited by the health care provider to participate.

Exclusion Criteria:

* < %35 Excess weight loss

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-07; Primary Completion 2012-01 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
plasma concentrations of representative hormones of hunger and satiety | 2 weeks

SECONDARY OUTCOMES:
surveying hunger/satiety and behavior changes. | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Francois Fritz, M.D., Principal Investigator — NYUSOM
Locations (1):
- NYUSOM, New York, New York, United States